CLINICAL TRIAL: NCT01651039
Title: A Phase II, Single-Center, Open-Label Study Of Oral Panobinostat (LBH589) When Administered In Combination With Lenalidomide And Weekly Dexamethasone In Patients With Multiple Myeloma
Brief Title: Phase II, Single-Center, Oral Panobinostat in Combination With Lenalidomide and Dexamethasone in Multiple Myeloma (MM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ajai Chari (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Ajai Chari, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-0469; CLBH589DUS85T
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma
Keywords: Panobinostat; Lenalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — Panobinostat; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panobinostat, Lenalidomide and Dexamethasone (Experimental): All patients will receive oral panobinostat, lenalidomide and dexamethasone as per protocol.
  Interventions: Drug: Panobinostat; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Panobinostat — Each cycle is 28 days. Panobinostat will be given 20 mg: Days 1,3,5,15,17,19.
  Other Names: LBH589
Drug: Lenalidomide — Each cycle is 28 days. Lenalidomide will be given 25 mg: Days 1-21.
  Other Names: Revlimid
Drug: Dexamethasone — Each cycle is 28 days. Dexamethasone will be given for patients 75 years old and younger a dose of 40 mg on Days 1, 8 and 15. Dexamethasone will be given for patients older than 75 years old, 20 mg on Days 1, 8 and 15.

SUMMARY:
The purpose of this clinical research study is to find out the effects of a drug called panobinostat (LBH589) when given to people like you with multiple myeloma in combination with the drugs lenalidomide and dexamethasone. The safety of this combination of drugs will also be studied. Your physical state, changes in the state of your multiple myeloma, and laboratory findings taken while on-study will help us decide if panobinostat combined with dexamethasone and lenalidomide is safe and effective.

This goal of this study therefore is to determine the activity of the combination of panobinostat thrice weekly every other week, lenalidomide, and weekly dexamethasone in a similar group of subjects. The doses of lenalidomide and dexamethasone will be that which is approved by the FDA for multiple myeloma and you will take each drug at a specific frequency over a 4 week (28 day) period. This period is called a "study cycle".

DETAILED DESCRIPTION:
The study drug, panobinostat, is made by Novartis Pharmaceuticals Corporation. Panobinostat has not yet been approved by the Food and Drug Administration (FDA) and thus is considered an experimental drug in this research study. Panobinostat is not available to you "on the market" (available for you to buy). It is only available in clinical trials for patients like you with your medical condition. Panobinostat is a drug that may slow down the growth of multiple myeloma or kill multiple myeloma cells by blocking certain enzymes (proteins produced by cells). Panobinostat has shown effects against cancers such as multiple myeloma in laboratory studies and in studies using animals; however, it is not known if this medicine will show the same activity in humans. As of 31st December 2009, a total of 1116 patients have already received treatment with panobinostat.

Unlike panobinostat, lenalidomide (Revlimid©) and dexamethasone are approved by the FDA and are already available for purchase on the US market. Clinical trials have shown that lenalidomide, especially taken with dexamethasone, produces positive clinical responses with manageable side effects when given to subjects with multiple myeloma.

In this study, subjects will take panobinostat capsules, lenalidomide, and dexamethasone all orally. The purpose of this combination is to interfere with the cancerous cells in multiple and different ways as each of these drugs acts differently on cancer cells. By combining the drugs and giving them at the same time, it might be possible to slow the progression of your disease, rather than if study drugs were given separately. Researchers have combined laboratory studies on animals with this drug combination and the combined effect has been shown to be worthwhile to justify clinical trials in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a history of symptomatic multiple myeloma according to the International Myeloma Working Group criteria (IMWG, 2003), as defined as the following three criteria:

   1. Clonal plasma cells >10% on bone marrow biopsy
   2. A monoclonal protein (paraprotein) in either serum or urine(except in cases of non-secretory myeloma)
   3. Evidence of end-organ damage felt related to the plasma cell disorder (related organ or tissue impairment, ROTI, commonly referred to by the acronym "CRAB"):

      * Hypercalcemia serum Ca ≥ 11.5 mg/dL or
      * Renal insufficiency attributable to myeloma. Serum creatinine > 2mg/dL
      * Anemia: Normochromic, normocytic with a hemoglobin value > 2g/dL below the lower limit of normal or a hemoglobin <10 g/dL
      * Bone lesions (lytic lesions, severe osteopenia or pathologic fractures
2. Patients must have received at least one prior line of therapy. For example; One prior line of therapy may consist of all predetermined components of induction followed by autologous stem cell transplantation and maintenance.
3. Patient has relapsed or relapsed/refractory MM.

   1. Relapsed is defined as the development of disease progression following the achievement of stable disease (SD) or better to the most recent anti-MM regimen.
   2. Refractory is defined as experiencing less than a partial response (PR) to or progressive disease (PD) within 6 months after completion of the most recent anti-MM regimen.
4. Patients must currently have measureable disease, as defined as:

   1. a. Serum M protein ≥ 1.0 g/dl (≥ 10 mg/l)
   2. Urine M protein ≥ 200 mg/24h
   3. Serum free light chain assay: involved FLC level ≥ 10mg/dl (≥ 100 mg/l) provided serum FLC ratio is abnormal
   4. If no monoclonal protein is detected (non-secretory disease), then > 30% monoclonal bone marrow plasma cells.
5. Patients must be suitable (according to their local product information) for treatment or re-treatment with lenalidomide & dexamethasone. Note: patients previously treated with lenalidomide & dexamethasone are eligible to participate in the trial.
6. Male or female adults ≥ 18 years old
7. ECOG Performance Status ≤ 2
8. Life expectancy > 12 weeks
9. Patients must have the following laboratory values:

   1. ANC ≥ 1.5 x 109/L for patients in whom < 50% of bone marrow nucleated cells are plasma cells; or an ANC > 1.0 x 109/Lfor patients in whom > 50% of bone marrow nucleated cells are plasma cells.
   2. Hemoglobin ≥ 9 g/dl
   3. Platelets ≥ 75x 109/L for patients in whom < 50% of bone marrow nucleated cells are plasma cells; or > 50 x 109/L for patients in whom > 50% of bone marrow nucleated cells are plasma cells.
   4. Calculated CrCl ≥ 50 mL/min (MDRD Formula)
   5. Hepatic:
   6. AST and ALT ≤ 2.5 x ULN,
   7. Serum bilirubin ≤ 1.5 x ULN
   8. Electrolytes:
   9. Serum potassium ≥ LLN,
   10. Total serum calcium [corrected for serum albumin] or ionized calcium ≥LLN
   11. Serum magnesium ≥ LLN
   12. Serum phosphorus ≥ LLN
   13. Normal thyroid function (TSH and free T4) (Clinically euthyroid patients are acceptable).
10. Able to sign informed consent and to comply with the protocol

Exclusion criteria

1. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment
2. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

   1. History or presence of sustained ventricular tachyarrhythmia. (Patients with a history of atrial arrhythmia are eligible but should be discussed with Novartis prior to enrollment)
   2. Any history of ventricular fibrillation or torsade de pointes
   3. Bradycardia defined as HR< 50 bpm. Patients with pacemakers are eligible if resting HR ≥ 50 bpm.
   4. Screening ECG with a QTc > 450 msec
   5. Right bundle branch block + left anterior hemiblock (bifascicular block)
   6. Patients with myocardial infarction or unstable angina ≤ 6 months prior to starting study drug
   7. Other clinically significant heart disease (e.g., CHF NY Heart Association class III or IV , uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
3. Impairment of GI function or GI disease that may significantly alter the absorption of panobinostat
4. Patients with diarrhea > CTCAE grade 2
5. Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
6. Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
7. Patients who have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is longer) and who have not recovered from side effects of those therapies.
8. Patients who have received either immunotherapy within < 8 weeks; chemotherapy within < 4 weeks; or radiation therapy to > 30% of marrow-bearing bone within < 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies.
9. Subject has received a cumulative dose of corticosteroids more than the equivalent of ≥ 140 mg of prednisone within the 2-week period before Cycle 1 Day 1.
10. Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
11. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not using an effective method of birth control. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential must have a negative serum pregnancy test within 24hrs of receiving the first dose of study medication.
12. Male patients whose sexual partners are WOCBP not using effective birth control
13. Patients with a prior malignancy with in the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
14. Patients with known positivity for human immunodeficiency virus (HIV) ) or hepatitis C; baseline testing for HIV and hepatitis C is not required
15. Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.
16. Patients with a history of Deep Vein Thrombosis or thromboembolism within < 6 months prior to starting study treatment
17. Patients for whom prophylactic anticoagulation therapy (eg. 325mg aspirin PO daily or warfarin (Coumadin®) 1-2 mg/day, or any other coumarin-derivative anticoagulants) is not an option.
18. Patients who have received allogeneic stem cell transplantation < 12 months prior to entering the study
19. Patients who have had prior allogeneic stem cell transplantation and show evidence of active graft-versus-host disease that requires immunosuppressive therapy.
20. All patients must agree to follow the requirements for lenalidomide counseling, pregnancy testing and birth control. For women of childbearing potential (WOCBP) this includes pregnancy testing prior to prescribing lenalidomide and to either commit to continued abstinence from heterosexual intercourse or begin acceptable methods of birth control for 28 days prior to prescribing lenalidomide, during therapy and for 28 days after the last dose of lenalidomide. WOCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a WOCBP even if they have had a successful vasectomy and must agree not to donate semen during study drug therapy and for a period of time after therapy. All patients must abstain from donating blood, agree not to share lenalidomide with others and be counseled about the risks of lenalidomide. See Appendix 2 requirements including the definition of WOCBP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajai Chari, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in July 2012 with enrollment from Sept 2012 to August 2015. 41 subjects signed consent (7 screened failed, 32 received study treatment, 5 non-evaluables). 27 out of the 32 subjects are evaluable.
Groups:
- Panobinostat, Lenalidomide and Dexamethasone: All patients will receive oral panobinostat, lenalidomide and dexamethasone as per protocol.
  Panobinostat, Lenalidomide and Dexamethasone: Each cycle is 28 days. Panobinostat will be given 20 mg: Days 1,3,5,15,17,19. Lenalidomide will be given 25 mg: Days 1-21. Dexamethasone will be given for patients 75 years old and younger a dose of 40 mg on Days 1, 8 and 15. Dexamethasone will be given for patients older than 75 years old, 20 mg on Days 1, 8 and 15.
Period: Overall Study
Arm/Group | Panobinostat, Lenalidomide and Dexamethasone
Started | 32
Completed | 2
Not Completed | 30
Not completed — Non-evaluables | 5
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1
Not completed — Progressive Disease | 22

BASELINE CHARACTERISTICS:
Population: 27 out of the 32 subjects are evaluable because the 5 patients either did not complete cycle 1, or enrolled but never dosed.
Arm/Group | Panobinostat, Lenalidomide and Dexamethasone
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 64 [51 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 16
Age >65 years [Count of Participants; unit: Participants] | 14
The Eastern Cooperative Oncology Group (ECOG) Performance [Count of Participants; unit: Participants] — ECOG measures level of functioning in terms of daily living abilities:
  0 - Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    0 | 16
    1 | 11
    2 | 0
ISS Staging [Count of Participants; unit: Participants] — The International Staging System (ISS) for Multiple Myeloma
  Stage 1 ß2-M < 3.5 mg/dL and albumin =3.5 g/dL
  Stage 2 Neither stage 1 nor stage 3
  Stage 3 ß2-M ≥ 5.5 mg/L
  Participants
    Stage 1 | 5
    Stage 2 | 5
    Stage 3 | 5
    missing | 12
Immunoglobulin subtype [Count of Participants; unit: Participants]
  IgG | 14
  IgA | 8
  IgM | 1
  None | 4
FISH [Count of Participants; unit: Participants]
  Normal | 2
  Any abnormality | 22
  Any high risk abnormality | 17
  del(17p) | 5
  chr1 amplification | 12
  t(4;14) | 4
  del(13q) | 5
  t(11;14) | 5
Median time since diagnosis [Median (Full Range); unit: years] | 4 [1.6 to 12.4]
Prior regimens [Median (Full Range); unit: years] — Number of years participant was on any prior regimens
  years | 3 [1 to 10]
Prior therapy [Median (Full Range); unit: regimens] — The number of prior treatments the participants had received prior to baseline visit
  regimens | 3 [1 to 10]
Prior Therapy, Exposed [Count of Participants; unit: Participants] — The number of participants that received any of the following chemo drugs
  Participants
    Dexamethasone | 27
    Thalidomide | 6
    Lenalidomide | 27
    Pomalidomide | 10
    Bortezomib | 27
    Carfilzomib | 8
    Autologous stem cell transplant | 20
Prior therapy, Refractory [Count of Participants; unit: Participants] — The number of participants that received any of the following chemo drugs and relapsed from it.
  Participants
    Dexamethasone | 19
    Thalidomide | 2
    Lenalidomide | 22
    Pomalidomide | 19
    Bortezomib | 14
    Carfilzomib | 7
Median cumulative duration of prior lenalidomide (len) months [Median (Full Range); unit: months] | 13 [4 to 20]
Prior len regimens [Median (Full Range); unit: regimens] | 1 [1 to 2]
Doses of lenalidomide at time of PD on len [Count of Participants; unit: Participants]
  25 | 7
  15 | 5
  10 | 7
  5 | 1
  unknown | 2
  Not Len Refractory Patients | 5
Progressed while on last len regimen [Count of Participants; unit: Participants] | 22
Len in most recent prior regimen [Count of Participants; unit: Participants] | 13
Pom in most recent prior regimen [Count of Participants; unit: Participants] | 3
Dex in most recent prior regimen [Count of Participants; unit: Participants] | 21
Dex in last len-containing regimen [Count of Participants; unit: Participants] | 23
Best response at last treatment [Count of Participants; unit: Participants]
  Complete response | 2
  Very Good Partial Response | 4
  Partial Response | 5
  Minimal Response | 9
  Stable Disease | 6
  Progressive disease | 1

OUTCOME MEASURES:

1. Primary Outcome: The Best Overall Response Rate (ORR)
Description: The primary endpoint will be the best overall response rate (ORR). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to 4 years
Measure: Count of Participants; unit: Participants
Groups:
- Panobinostat, Lenalidomide and Dexamethasone: All patients received oral panobinostat, lenalidomide and dexamethasone as per protocol
Arm/Group | Panobinostat, Lenalidomide and Dexamethasone
Number analyzed (Participants) | 27
Participants | 11

2. Primary Outcome: Overall Response Rate for Len Refractory Patients
Description: The primary endpoint will be the best overall response rate (ORR)
Time Frame: up to 4 years
Population: Only Len Refractory Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat, Lenalidomide and Dexamethasone
Number analyzed (Participants) | 22
Participants | 8

3. Secondary Outcome: Response Rates
Description: Response Rates evaluated using the International Uniform Response Criteria the International Myeloma Working Group (2003).
  CR-Negative immunofixation on the serum and urine and Disappearance of any soft tissue plasmacytomas and 5% plasma cells in bone marrow VGPR-Serum and urine M-component detectable by immunofixation but not on electrophoresis or 90 or greater reduction in serum M-component plus urine M-component <100 mg per 24 h PR-50% reduction of serum M-protein and reduction in 24-h urinary M-protein by 90% or to <200 mg per 24 h MR-≥ 25% but < 49% reduction of serum M protein and reduction in 24 hour urine M protein by 50 - 89%, which still exceeds 200 mg/24hrs. In addition; if present at baseline, 25-49% reduction in the size of soft tissue plasmacytomas also required No increase in size or number of lytic bone lesions.
  SD-Not meeting criteria for CR, VGPR, PR or progressive disease PD-Laboratory or Biochemical Relapse increase of 25% from baseline
Time Frame: up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat, Lenalidomide and Dexamethasone
Number analyzed (Participants) | 27
Participants
  Complete Response (CR) | 2
  Very Good Partial Response (VGPR) | 4
  Partial Response (PR) | 5
  Minimal Response (MR) | 9
  Stable Disease (SD) | 6
  Progressive Disease (PD) | 1

4. Secondary Outcome: Response Rates for Len Refractory Patients
Description: as for outcome 3
Time Frame: up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat, Lenalidomide and Dexamethasone
Number analyzed (Participants) | 22
Participants
  Complete Response | 1
  Very Good Partial Response | 4
  Partial Response | 3
  Minimal Response | 7
  Stable Disease | 6
  Progressive Disease | 1

5. Secondary Outcome: Clinical Benefit Rate
Description: The number of response rates in participants that have achieved MR, PR, VGPR, CR
Time Frame: up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat, Lenalidomide and Dexamethasone
Number analyzed (Participants) | 27
Participants | 20

6. Secondary Outcome: Clinical Benefit Rate for Len Refractory Patients
Description: The number of response rates in Lens Refractory participants that have achieved MR, PR, VGPR, CR
Time Frame: up to 4 years
Population: Only Len Refractory Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat, Lenalidomide and Dexamethasone
Number analyzed (Participants) | 22
Participants | 15

7. Secondary Outcome: Disease Control Rate
Description: The number of response rates participants with SD, MR, PR, VGPR, or CR
Time Frame: up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat, Lenalidomide and Dexamethasone
Number analyzed (Participants) | 27
Participants | 26

8. Secondary Outcome: Disease Control Rate for Lens Refractory Rate
Description: The number of response rates in Len refractory participants with SD, MR, PR, VGPR, or CR
Time Frame: up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat, Lenalidomide and Dexamethasone
Number analyzed (Participants) | 22
Participants | 21

ADVERSE EVENTS:
Description: Adverse events collected for all subjects who signed consent
Groups:
- All Subjects: Adverse events collected for all subjects who signed consent.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 1/41
Serious Adverse Events (participants affected / at risk) | 14/41
Other Adverse Events (participants affected / at risk) | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=41)
Cardiac Catherization (Cardiac disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Ehrlichiosis Babesiosis (Infections and infestations) | 1 (1)
Failure to thrive (General disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Lap low Anterior Surgery (Surgical and medical procedures) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary Embolism (Blood and lymphatic system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Shortness of breath (General disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=41)
Abdominal Pain (Gastrointestinal disorders) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Acute GI upset (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
acute renal insufficiency (Renal and urinary disorders) | 1 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Alanine Aminotransferase (Metabolism and nutrition disorders) | 2 (2)
Allergic rhinitis (General disorders) | 1 (1)
Alk phos elevation (Metabolism and nutrition disorders) | 1 (1)
ALT elevation (Metabolism and nutrition disorders) | 1 (2)
ALT increased (Metabolism and nutrition disorders) | 1 (2)
Altered smell (General disorders) | 1 (1)
Altered taste (General disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 18 (56)
Anorexia (General disorders) | 7 (8)
anorexia intermittent (General disorders) | 1 (1)
Atypical Chest Pain (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Balance issue (Nervous system disorders) | 1 (1)
Bilateral knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral lower extremity cramps (Musculoskeletal and connective tissue disorders) | 2 (2)
Bilateral leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral lower extremity swelling (Vascular disorders) | 3 (3)
bilateral submandibular lymph node pain (Blood and lymphatic system disorders) | 1 (1)
bilirubin increase (Hepatobiliary disorders) | 3 (5)
Bleeding gums (General disorders) | 1 (1)
Bloating (General disorders) | 2 (2)
Blood in stool (Gastrointestinal disorders) | 1 (1)
Blurry vision (Eye disorders) | 1 (1)
Body aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain - Right wrist (Musculoskeletal and connective tissue disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (2)
Bruising (Blood and lymphatic system disorders) | 1 (1)
Bruising (right abd) (Blood and lymphatic system disorders) | 1 (1)
Burning would right foot (General disorders) | 1 (1)
C. Difficile (Infections and infestations) | 1 (1)
Cataracts in both eyes (Eye disorders) | 1 (1)
C3-C4 compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Cheek flushing (General disorders) | 1 (1)
Cheek pain (General disorders) | 1 (2)
Cheiilitis (Skin and subcutaneous tissue disorders) | 1 (1)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Chest Pain Intermittent (General disorders) | 1 (1)
Chest tightness (General disorders) | 1 (1)
Chills (General disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1) — T wave inversion
Confusion (Nervous system disorders) | 1 (1)
Congestion (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 13 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (16)
Cough/cold (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cramping (Musculoskeletal and connective tissue disorders) | 1 (1)
Cramps on both legs (Musculoskeletal and connective tissue disorders) | 1 (1)
Creatinine increase (Hepatobiliary disorders) | 2 (2)
decreased appetite (Gastrointestinal disorders) | 1 (1)
Dental abscess (Infections and infestations) | 1 (1)
Depression (Psychiatric disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 16 (29)
Diarrhea intermittent (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7)
Dizziness intermittent (Nervous system disorders) | 1 (1)
Cough, dry (General disorders) | 1 (1)
Dry eyes (Eye disorders) | 1 (1)
Dry mouth (General disorders) | 2 (2)
DVT left leg (Blood and lymphatic system disorders) | 1 (1)
DVT right leg (Blood and lymphatic system disorders) | 1 (1)
Dyspnea on exertion (General disorders) | 2 (2)
Dyspepsia (General disorders) | 2 (4)
Dyspnea (General disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Edema (Blood and lymphatic system disorders) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 2 (3)
Facial swellinig (General disorders) | 1 (1)
Fall (General disorders) | 2 (3)
Fatigue (General disorders) | 23 (44)
Fatigue (post dex) (General disorders) | 1 (3)
Fever (General disorders) | 7 (14)
Fistula (Gastrointestinal disorders) | 1 (1) — colon/bladder
Flank/lats discomfort (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Foam in urine (Renal and urinary disorders) | 2 (2)
forehead bumps (General disorders) | 1 (1)
Fungal rash (Infections and infestations) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 (4)
GI symptoms (Gastrointestinal disorders) | 1 (1)
Gum irritation (General disorders) | 1 (1)
Hand cramps (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (General disorders) | 5 (7)
Headache, intermittent (General disorders) | 2 (2)
Hematoma (Blood and lymphatic system disorders) | 1 (1) — right forearm
Hematuria (Renal and urinary disorders) | 2 (2)
Hemorrhoid pain (Gastrointestinal disorders) | 1 (1)
Hiccups (General disorders) | 1 (1)
Hoarse voice (General disorders) | 2 (2)
Hoarseness (General disorders) | 2 (2)
hot flashes (General disorders) | 1 (1) — post dex
hyperbilirubinemia (Metabolism and nutrition disorders) | 2 (2)
hypercalcemia (Metabolism and nutrition disorders) | 3 (6)
hyperglycemia (Metabolism and nutrition disorders) | 2 (7)
hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2)
hyperpigmentation of soles (General disorders) | 1 (1)
hypersalivation (General disorders) | 1 (1)
hypertension (Cardiac disorders) | 3 (7)
hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
hypocalcemia (Metabolism and nutrition disorders) | 1 (4)
hypoguesia (General disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 7 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
hypomagnesia (Metabolism and nutrition disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (7)
hypophosphorous (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (4)
Hypoxia (General disorders) | 1 (1)
increased blood sugar (Metabolism and nutrition disorders) | 1 (1)
increased creatinine (Metabolism and nutrition disorders) | 1 (1)
increased gas (General disorders) | 1 (1)
increased phosphorus (General disorders) | 1 (3)
increased thirst (General disorders) | 1 (1)
infection (Infections and infestations) | 1 (1)
influenza (Infections and infestations) | 1 (1)
insomnia (General disorders) | 10 (12)
insomnia (post dex) (General disorders) | 1 (1)
intermittent diarrhea (Gastrointestinal disorders) | 1 (1)
intermittent dry cough (General disorders) | 1 (1)
intermittent headache (General disorders) | 1 (1)
intermittent heartburn (General disorders) | 1 (1)
intermittent itching (Skin and subcutaneous tissue disorders) | 1 (1)
jaw pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Jitters (with dex) (General disorders) | 1 (2)
L rib pain (Musculoskeletal and connective tissue disorders) | 2 (2)
L Upper Leg Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
LE edema (General disorders) | 2 (7)
LE weakness (General disorders) | 1 (1)
Left ankle edema (General disorders) | 1 (1)
Left lower extremities deep vein thrombosis (Blood and lymphatic system disorders) | 1 (1)
Left sternal pain (intermittent) (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg cramps (General disorders) | 4 (4)
leukocyte count decreased (Blood and lymphatic system disorders) | 7 (14)
leukopenia (Blood and lymphatic system disorders) | 4 (8)
localized edema (General disorders) | 1 (1)
loose stools (Gastrointestinal disorders) | 1 (1)
Low magnesium (Metabolism and nutrition disorders) | 2 (2)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Lower extremity edema (General disorders) | 1 (1) — L>R
Lymphopenia (Blood and lymphatic system disorders) | 7 (25)
Malaise (General disorders) | 2 (2)
Mid back bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Mid-back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Mildly elevated phosphorus (Metabolism and nutrition disorders) | 1 (1)
Minor congestion dry cough (General disorders) | 1 (1)
Mood irritability (General disorders) | 1 (1)
Mood Swings/Confusion (General disorders) | 1 (1)
Mouth sore (General disorders) | 2 (2)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nasal congestion (General disorders) | 1 (1)
Nausea (General disorders) | 11 (16)
Nausea intermittent (General disorders) | 1 (1)
Nausea/vomiting (General disorders) | 1 (1)
Neck numbness (General disorders) | 1 (1)
Neck pain (General disorders) | 2 (2)
Neuropathy (General disorders) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 26 (176)
Nightsweats (General disorders) | 1 (1)
Nose bleeding (General disorders) | 1 (1)
Optic nerve damage (Eye disorders) | 1 (1)
Oral Thrush (Infections and infestations) | 1 (1)
Pain at the base of skull (General disorders) | 1 (1)
Pain on upper extremities (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Paronchytis (Infections and infestations) | 1 (1)
Pedal Edema (General disorders) | 2 (2)
Peripheral Neuropathy (General disorders) | 1 (1)
Peripheral Neuropathy Bilateral (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Pneumonia (SOB) (Infections and infestations) | 1 (2)
Poor appetite (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes